CLINICAL TRIAL: NCT06144593
Title: The Metabolic Impact of Intermittent Carbohydrate Restriction in Individuals With Type 2 Diabetes
Acronym: INTERCARB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Danish Research Centre for Magnetic Resonance (Other)
Responsible Party: Principal Investigator, Kirstine Nyvold Bojsen-Moeller, MD, PhD, Associate Professor, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: INTERCARB - H-23043085
Record Dates: First submitted 2023-09-29; First posted 2023-11-22 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity; Non-Alcoholic Fatty Liver Disease; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Dietary intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent carbohydrate restriction (Experimental): Four weeks of intermittent carbohydrate restriction: a dietary regime alternating between two days of restricting carbohydrate intake to 70-90 grams, while energy intake is ad libitum, from fat- and protein-containing foods, and two days of non-restricted diet.
  Interventions: Other: Dietary macronutrient composition
- Control arm (No Intervention): Four weeks of free-living with no dietary restrictions.

INTERVENTIONS:
Other: Dietary macronutrient composition — Intermittent carbohydrate restriction
  Arms: Intermittent carbohydrate restriction

SUMMARY:
The primary aim of this randomized cross-over intervention study is to investigate the effect of four weeks of intermittent carbohydrate restriction (alternating between two days of normal dietary intake and two days of carbohydrate restriction to 70-90 grams) on 24-hour average sensor glucose in individuals with type 2 diabetes compared with a four-week control period with normal dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* 35-75 years old
* BMI >27 kg/m2
* Known type 2 diabetes in stable glucose lowering therapy (for three months) or with HbA1c >48 mmol/mol if no glucose lowering therapy

Exclusion Criteria:

* Anemia (hemoglobin <8 mmol/L for men and <7 mmol/L for women)
* TSH outside reference range
* Treatment with insulin, sulfonylurea, or SGLT2-inhibitors
* Treatment with systemic corticosteroids
* HbA1c >70 mmol/mol
* eGFR <60 ml/min/1.73 m2
* Contraindications for MR-scan: abdominal height exceed limitations of the MR-scanner, pacemaker or other electronic device implanted, implanted metal devices, severe claustrophobia
* Food allergies (including lactose and gluten intolerance)
* Vegetarian/vegan diet or following of specific dietary plans
* Alcohol consumptions >84/168 g/week (women/men)
* Strenuous activity level > 120 minutes per week
* Weight loss (>5 kg) within the last three months or previous bariatric surgery
* High risk of fibrosis of the liver (estimated by FIB4 score > 3.25)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
24-hour average sensor glucose | 24-hour average sensor glucose is measured as the average of eight consecutive days (starting from two days post sensor mounting) from the intermittent carbohydrate restriction period and the corresponding days of the control period (i.e. days 17-24).
  A patient-blinded continuous glucose monitoring (CGM) is worn during the last two weeks of both the intervention and control period.

SECONDARY OUTCOMES:
Liver triacylglycerol content | day 30 adjusted for baseline
  Liver TG content will be measured by 1H-Magnetic Resonance Spectroscopy (MRS) on the day before and the day after the 4-week dietary intervention (i.e. day 0 and day 30) and on the day before and the day after the 4-week control period (i.e. day 0 and day 30).
Fasting plasma concentrations of triacylglycerols | day 30 adjusted for baseline
  Fasting plasma concentrations of triacylglycerols measured on the day before and the day after the 4-week dietary intervention (i.e. day 0 and day 30) and on the day before and the day after the 4-week control period (i.e. day 0 and day 30).

OTHER OUTCOMES:
Explorative outcomes - Questionnaires on quality of life | day 30
  Participants will complete the questionnaires 'Problem Areas In Diabetes' & 'World Health Organisation-Five Well-Being Index'.
Explorative outcomes - Qualitative evaluation to assess feasibility of the dietary strategy | day 30
  A semi-structured evaluation interview to assess social context, eating practices, compliance to, and feasibility and acceptability of the intermittent carbohydrate restriction regime will be carried out.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Hvidovre Hospital, Hvidovre, Denmark